CLINICAL TRIAL: NCT00527449
Title: Neoadjuvant Chemotherapy With 3x Epirubicin/Docetaxel Followed by 3x Carboplatin/Docetaxel in Patients With Primary Breast Cancer
Brief Title: Neoadjuvant Chemotherapy of Primary Breast Cancer With Epirubicin/Docetaxel and Carboplatin/Docetaxel
Acronym: ETCat01
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Klinikum Weissenfels (Other)
Responsible Party: Dieter Lampe, Dr. med., Klinikum Weissenfels
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3305000
Record Dates: First submitted 2007-09-07; First posted 2007-09-10 (Estimated); Last update posted 2010-01-15 (Estimated); Status verified 2010-01

CONDITIONS: Primary Breast Cancer
MeSH Terms: interventions — Epirubicin; Carboplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Epirubicin, Carboplatin, Docetaxel — 75 mg/m² Docetaxel (60 minutes i.v.) and 90 mg/m² Epirubicin (10-15 min i.v.) on day 1, 22, 42. After these 3 cycles 75 mg/m² Docetaxel (60 minutes i.v.) and Carboplatin AUC 5 (30 min i. v.) on day 63, 84, 105.

SUMMARY:
The purpose of this study is to optimize results in neoadjuvant chemotherapy of local advanced primary breast cancer. Therefore patients become first 3 cycles of Epirubicin/Docetaxel followed by 3x Carboplatin/Docetaxel.

DETAILED DESCRIPTION:
Most of the women who are diagnosed with breast cancer are in the situation that an operation is possible. Using a neoadjuvant therapy the rate of breast-conserving surgery can be extended and tumor cell proliferation may be inhibited. Further the neoadjuvant chemotherapy is an in-vivo-activity-test for the used drugs. Epirubicin, Docetaxel and Carboplatin have shown antineoplastic activity against solid cancer alone and in combination.

Using two different combinations of these three drugs, first 3 cycles Epirubicin/Docetaxel and then changing to Carboplatin/Docetaxel for 3 further cycles it is assumed that the results of the therapy will improve. Main criterion is the determination of pCR, second criteria are the rate of breast-conserving surgery, tumor response and therapy-dependent toxicities.

ELIGIBILITY:
Inclusion Criteria:

* histologically assured breast cancer
* age >= 18 years
* bone marrow function: neutrophils >= 1.5x109/l, platelets >= 100x109/l, hemoglobin >=6.2 mmol/l
* sufficient renal and liver function
* ECOG 0-2
* written informed consent

Exclusion Criteria:

* pregnant or nursing women
* distant metastases
* T2-Tumour < 3cm and G1
* existing motoric or sensoric neurotoxicity > Grade 2
* known hypersensitivity against Epirubicin or other anthracycline or against Carboplatin or other platin derivatives or against Docetaxel or against substances in the preparing solutions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-05; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Determining pathologic complete remission under study treatment | 28 days after last administration of chemotherapy

SECONDARY OUTCOMES:
Rate of breast conserving operations | 28 days after administration of last chemotherapy
Response to treatment | 28 days after last administration of chemotherapy
Determining the therapy associated toxicity | 28 days after last administration of chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Lampe, Dr. med., Principal Investigator — Asklepios Krankenhaus Weissenfels
Locations (3):
- Germany (3):
  - Krankenhaus St. Elisabeth u. St. Barbara, Halle, Saxony-Anhalt
  - Klinikum Marienstift, Magdeburg, Saxony-Anhalt
  - Asklepios Krankenhaus Weissenfels, Weißenfels, Saxony-Anhalt